CLINICAL TRIAL: NCT05156216
Title: Comparative Effect of Two Educational Videos for People With Knee Osteoarthritis - Disease and Impairment Discourse Versus Empowerment and Participatory Discourse: vidEO - An Online Randomised Controlled Trial
Brief Title: Comparative Effect of Two Educational Videos for People With Knee Osteoarthritis (vidEO)
Acronym: vidEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT21063; U1111-1269-6143 (Other: Universal Trial Number - World Health Organization)
Record Dates: First submitted 2021-11-10; First posted 2021-12-14 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Knee Osteoarthritis; Patient Empowerment
Keywords: knee osteoarthritis; patient education; health information; empowerment discourse; video; randomised controlled trial
MeSH Terms: conditions — Osteoarthritis, Knee; Patient Participation | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to one of two groups (1:1) using the randomiser function in Qualtrics (set to 'evenly present elements').
Who Masked: Participant, Outcomes Assessor
Masking Description: Limited disclosure will be used to blind participants and thereby reduce bias in responses since participants are also the assessors as all outcome measurements are self-reported. Participants will simply be informed that the trial aim is to assess knee OA educational videos. The investigators will not disclose details about how the educational content/presentation of the two videos differ, nor the hypotheses of the study. The biostatistician who performs the data analysis will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental video (Experimental): Knee OA educational video based on an empowerment discourse delivered online and embedded within the survey.
  Interventions: Other: Patient education
- Control video (Active Comparator): Knee OA educational video based on a disease and impairment discourse delivered online and embedded within the survey.
  Interventions: Other: Patient education

INTERVENTIONS:
Other: Patient education — Knowledge and beliefs about the condition and its management influences patient behavioural intentions, including treatment choices. Thus, patient education may play an important role in facilitating desirable behaviours with the aim of education being to develop accurate beliefs about treatment options and empower people to choose wisely for their current needs and circumstances.
  Other Names: Health information

SUMMARY:
Education is an important part of knee osteoarthritis management. The aim of education is to help people with knee osteoarthritis make the best choices for them in terms of their treatment and lifestyle behaviours. Traditional education that describes the condition simplistically in terms of the joint damage and describes the cause of osteoarthritis solely with respect to loading through the joint can lead to activity avoidance and pessimism about the future progression of symptoms. An alternative is to provide the information about knee osteoarthritis management with the aim of giving hope for the future and building motivation and confidence to be physically active. This study will compare two educational videos that cover the same topics but with a contrasting 'discourse'. The experimental video has an 'empowerment and participatory' discourse, while the comparator or control video has a typical 'disease and impairment' discourse. The experimental video minimises mention of joint damage and instead corrects misconceptions about knee osteoarthritis, addresses common barriers to physical activity and incorporates behaviour change techniques such as social learning and modelling of desired behaviours. In this randomised controlled trial, people who report a history of knee problems consistent with knee osteoarthritis will complete questionnaires to determine their self-efficacy for managing knee osteoarthritis pain and their fear of movement. The participants will also be asked about their expectations for the future, their level of motivation to be physically active, and their knowledge about knee osteoarthritis. Participants will then be allocated one of the videos and asked to watch it before repeating the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* live in Australia;
* are aged 45 years or over;
* have experienced activity-related knee pain during the past 3 months or have been told by a health professional that they have knee OA, ; and
* are able to easily understand verbal and written English language.

Exclusion Criteria:

* have had a hip or knee joint replacement;
* are scheduled/referred to see an orthopaedic surgeon or are already on a waiting list for hip or knee joint replacement;
* have any type of systemic arthritis (e.g. rheumatoid arthritis, gout), or have morning stiffness that lasts longer than 30 minutes;
* have a health condition that makes them unable to walk (since it will be difficult for people who cannot walk to follow the recommendations made in either video);
* have seen a health professional for their knee pain during the previous six months

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Self-efficacy for managing pain from osteoarthritis | Immediately post intervention
  Self-efficacy is considered fundamental for effective chronic disease self-management and greater self-efficacy is related to higher physical activity levels in people with OA. Self-efficacy will be measured with the Arthritis Self-Efficacy Scale (ASES) (pain subscale). Range 0-10, higher scores mean better self-efficacy.
Kinesiophobia | Immediately post intervention
  Kinesiophobia is the fear that movement will exacerbate pain. According to the fear-avoidance model, fear is worsened by heightened negative emotion and hypervigilance to symptoms. Kinesiophobia will be measured with the Brief Fear of Movement Scale for Osteoarthritis (BFMS). Range 6-24, lower scores mean better outcome.

SECONDARY OUTCOMES:
Expectations about their knee OA prognosis and benefit from physical activity | Immediately post intervention
  The Credibility/Expectations Questionnaire, which was designed to measure expectation of benefit from therapy, was adapted to measure expectations about their knee OA prognosis and the perceived effect of physical activity.There are two parts, Part 1: range 3-27, higher scores better. Part 2: range 2-18, higher scores better.
Importance of physical activity | Immediately post intervention
  Perceived importance of being physically active will be measured through rating the level of agreement with four statements. Likert scaling with 5 response options. Responses averaged so scores range 1-5. Two items reverse scored so that high scores indicate better.
Knee OA knowledge | Immediately post intervention
  Knowledge and beliefs about knee OA will be measured using the Knee Osteoarthritis Knowledge Scale (KOAKS). This scale has established content validity and is currently being examined for other psychometric properties. It currently has 15 items and scores range from 15-75 with higher scores indicated better knowledge, however, some items may be removed once reliability study is published.
Perceived change in feelings about having knee OA | Immediately post intervention
  Post-intervention change in feelings about having knee OA (specifically "How much have your feelings of hope for the future changed since watching the video?"), will be rated using a Likert scale with 5 response options. Responses will be dichotomised with participants indicating they are "somewhat more" or "much more" classified as 'more hopeful'. All other respondents classified as 'not more hopeful'.
Perceived personal likelihood of ever needing knee surgery | Immediately post intervention
  Perceived personal chance of ever having surgery will be measured using 5 level Likert scale from very unlikely to very likely. Scores range 1-5 with lower scores being considered better.
Motivation to be physically active | Immediately post intervention
  Motivation to be physically active will be determined by asking participants to rate 'How motivated are you to be physically active (e.g., walk, run, swim, cycle, dance, exercise, etc) even when you are feeling knee pain?', on a scale from 0 (not at all motivated) to 10 (very motivated). This question is drawn from the Information-Motivation-Behavioural skills model of behaviour change, which explains that having the motivation to change is an essential determinant of behaviour that is independent of both knowledge and behavioural skills. Range 0-10 with higher scores indicating greater motivation.

OTHER OUTCOMES:
Novelty check | Immediately post intervention
  Have you seen the video before? Yes/no
Fidelity check | Immediately post intervention
  How many times did you watch the video before completing this questionnaire? 0 = Did not watch the video or only watched part of the video
  1. = Watched it once through to the end
  2. = Watched it more than once through to the end
Satisfaction with the video education | Immediately post intervention
  How satisfied are you that the video helped meet your current needs for information about knee osteoarthritis? Single item Likert scale with 5 response options. Responses dichotomised to those indicating they are "moderately satisfied" or "very satisfied" classified as satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Thorlene Egerton, PhD, Principal Investigator — University of Melbourne
Locations (1):
- The University of Melbourne, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Egerton T, Bennell KL, McManus F, Lamb KE, Hinman RS. Comparative effect of two educational videos on self-efficacy and kinesiophobia in people with knee osteoarthritis: an online randomised controlled trial. Osteoarthritis Cartilage. 2022 Oct;30(10):1398-1410. doi: 10.1016/j.joca.2022.05.010. Epub 2022 Jun 22. PMID 35750241